CLINICAL TRIAL: NCT01659515
Title: Arbekacin Treatment of Adult Patients With Infections Caused by Multidrug-resistant Bacteria
Status: No longer available | Type: Expanded Access
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Meiji Seika Pharma Co., Ltd. (Industry); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: S-11-0001
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infection Due to Resistant Organism
MeSH Terms: interventions — arbekacin

INTERVENTIONS:
Drug: Arbekacin Sulfate — Intravenous arbekacin in a total daily dose of 5-7 mg/kg
  Other Names: Arbekacin; Habekacin

SUMMARY:
Arbekacin for the use of infection caused by multidrug-resistant organisms

DETAILED DESCRIPTION:
The primary purpose of this protocol is to make arbekacin available for treatment of patients with infections caused by multidrug-resistant organisms when treatment with other antibiotics cannot be used due to unavailability, intolerance, contraindications, or treatment non-response.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is military health care beneficiary at least 18 years of age;
2. Subject is a Walter Reed National Military Medical Center patient deemed by the primary medical or surgical team as having a bacterial infection of the respiratory tract, bloodstream, skin, soft tissue, bone, or genitourinary tract;
3. Subject is allergic to or intolerant of antibiotics to which the infective organism is susceptible; Or The use of antibiotics to which the subject's infective organism is susceptible is contraindicated; Or

   Subject's infective organism isolate is a multidrug-resistant (MDR) bacterium defined as any of the following:
   * Gram-negative bacterium that is non-susceptible to all index antibiotics within 3 or more of 6 antibiotic classes including aminoglycosides (amikacin, gentamicin, tobramycin), beta-lactam/beta-lactam inhibitor combinations (piperacillin-tazobactam, amoxicillin-clavulanate), carbapenems (imipenem, ertapenem), fluoroquinolones (ciprofloxacin, levofloxacin), cephalosporins (ceftazidime, cefepime, ceftriaxone), and sulbactam (ampicillin-sulbactam);
   * Extended Spectrum β-lactamase (ESBL) producing Gram-negative bacterium;
   * Carbapenemase resistant Enterobacteriaceae;
   * Cephalosporin resistant Klebsiella species;
   * Methicillin-resistant Staphylococcus aureus (MRSA);
   * Vancomycin resistant Enterococcus species;
   * Staphylococcus aureus that is non-susceptible to vancomycin.
4. Subject's infective organism is inhibited in vitro by arbekacin at a concentration ≤ 4 μg/mL;
5. Subject is able to give written or witnessed verbal informed consent [An exception from the general requirements for informed consent can be made based upon the criteria specified in 21 Code of Federal Regulations 50.23 (a and c)];
6. Subject has adequate venous access for intravenous administration of arbekacin.
7. Sexually active females, unless surgically sterile or at least 1 year post-menopausal, must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner, or sterile sexual partner) for at least 30 days prior to receipt of arbekacin and must agree to continue using such precaution for at least 30 days after last dose of arbekacin; the subject must also have a negative pregnancy test within 24 hours prior to initial dose of arbekacin.

Exclusion Criteria:

1. Subject has a history of allergy or serious adverse reaction to aminoglycoside antibiotics;
2. Subject is currently participating in another investigational new drug study.
3. Subject has a positive serum pregnancy test or is breast feeding.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapor, MD, PhD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed National Military Medical Center (WRNMMC), Bethesda, Maryland, United States